CLINICAL TRIAL: NCT00562770
Title: Open Label, Phase II Randomized Study of Oral Valganciclovir Versus Valacyclovir for Prophylaxis of Cytomegalovirus Reactivation in Patients Receiving Alemtuzumab (Campath).
Brief Title: Oral Valganciclovir Versus Valacyclovir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID02-666
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Lymphocytic Leukemia; Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — Valganciclovir; Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Valacyclovir
  Interventions: Drug: Valacyclovir
- 2 (Active Comparator): Valganciclovir
  Interventions: Drug: Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir — 900 mg (two 450 mg capsules) po QD during therapy and for 2 months post alemtuzumab initiation.
  Other Names: Valcyte
  Arms: 2
Drug: Valacyclovir — 500 mg po QD during therapy and for 2 months post alemtuzumab initiation.
  Other Names: Valtrex
  Arms: 1

SUMMARY:
To determine if the rate of cytomegalovirus reactivation during treatment with alemtuzumab (Campath) is reduced by the use of valganciclovir prophylaxis.

DETAILED DESCRIPTION:
Researchers will study the effectiveness of valganciclovir to help prevent cytomegalovirus infections in patients receiving alemtuzumab. Since alemtuzumab eliminates T-cells, which are the body's usual defense against viruses, patients taking alemtuzumab have an increased risk of developing CMV.

Before treatment, you will have a physical exam. You will also have around 3-4 tablespoons of blood drawn for routine tests and for tests to see if you have ever been exposed to CMV.

You will be randomly assigned (as in the toss of a coin) to one of two treatment groups. Participants in one group will be given treatment with valganciclovir. Participants in the other group will be given treatment with valacyclovir. This drug protects against herpes infections but not CMV.

If you are assigned to the group that will receive valganciclovir, you will take valganciclovir by mouth once a day starting of your first day of alemtuzumab therapy. You will continue to take valganciclovir for 2 months after the end of alemtuzumab therapy.

If you are assigned to the group that will receive valacyclovir, you will take valacyclovir by mouth once a day starting of your first day of alemtuzumab therapy. You will continue to take valacyclovir for 2 months after the end of alemtuzumab therapy.

Every 2 weeks while you are receiving alemtuzumab (usually 4-12 weeks)you will have a repeat blood test to look for CMV.

Your participation in this study will last for a maximum of 5 months.

This is an investigational study. Both valganciclovir and valacyclovir are FDA approved and commercially available. However, the use of valganciclovir for this study is experimental. valganciclovir will be provided free of charge during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving alemtuzumab
* Age > 15
* Signed informed consent form

Exclusion Criteria:

* Active cytomegalovirus disease or infection. Asymptomatic patients with positive CMV pp65 antigenemia will not be excluded.
* Patients with a creatinine clearance of < 10 ml/min as calculated via the Cockcroft-Gault equation.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-09; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
CBC, platelet and differential. BUN, creatinine, total bilirubin, alkaline phosphatase, LDH, SGPT | CBC, platelet and differential 2 weeks +/- 3 days for 8 weeks, and every 4 weeks +/- 3 days during the remainder of therapy. BUN, creatinine, total bilirubin, alkaline phosphatase, LDH, SGPT every 4 weeks +/- 3 days.

SECONDARY OUTCOMES:
CMV antigenemia | CMV antigenemia every 2 weeks +/- 3 days for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan O'Brien, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] O'Brien S, Ravandi F, Riehl T, Wierda W, Huang X, Tarrand J, O'Neal B, Kantarjian H, Keating M. Valganciclovir prevents cytomegalovirus reactivation in patients receiving alemtuzumab-based therapy. Blood. 2008 Feb 15;111(4):1816-9. doi: 10.1182/blood-2007-03-080010. Epub 2007 Nov 26. PMID 18039954
- See also: M.D. Anderson's Website — http://www.mdanderson.org